CLINICAL TRIAL: NCT05415501
Title: Structural Priming as a Treatment Component in Aphasia
Brief Title: Sentence Production Training in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Temple University (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ji Yeon Lee, Associate Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-659
Record Dates: First submitted 2022-05-16; First posted 2022-06-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Aphasia
Keywords: aphasia training; aphasia treatment; sentences; grammar
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Structural priming training (Experimental): Participants will be enrolled in 3 sessions of structural priming training (for experiment 1-3) or up to 15 treatment sessions (for experiment 4). Each session will be about 2 hour long, consisting of a set of tasks, including repeating, making, and remembering various types of sentences. In experiment 1-3, each participant will receive two different experimental priming conditions that are being compared within each session. In experiment 4, participants will receive a structural priming treatment in a single-subject design.
  Interventions: Behavioral: Sentence training

INTERVENTIONS:
Behavioral: Sentence training — Participants will be trained to read, make, and recall sentences during each session.

SUMMARY:
This project focuses on developing a novel treatment for sentence production and comprehension in aphasia, using implicit priming. First set of experiments will aim examine which learning conditions are most effective in creating maximal training gains. Then, in a later study, the investigators will develop and test the efficacy of a novel treatment study based on findings from the first set of the studies.

DETAILED DESCRIPTION:
Over five years, the investigators will conduct a series of studies to develop a novel intervention strategy for improving sentence production and comprehension in persons with aphasia. Specifically, the investigators will use implicit learning of grammar as a novel facilitator for language recovery in aphasia. The planned studies seek to test the hypothesis that implicit learning alters the central language system in PWA, creating lasting and generalized improvements in both sentence production and comprehension. Aim 1 will determine the extent to which different learning conditions modulate immediate and long-term improvement in sentence production. The investigators integrate multiple theories of language learning and apply them to make predictions about the trajectory of priming-induced learning in PWA. In Aim 2, using a set of eyetracking and sentence comprehension tasks, it will be investigated whether the effects of priming in production generalize to off-line (accuracy) and on-line (eye fixations) sentence comprehension and determine which learning conditions result in greater cross-modality generalization. In Aim 3, the investigators will develop and establish Phase I efficacy data of an implicit priming treatment, incorporating the crucial learning conditions supporting maximal retention from Aims 1 and 2. The project will recruit both individuals with aphasia and without aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with post-stroke aphasia
* At least 6 months post-onset of eft hemisphere stroke
* Native speaker of English
* Normal or corrected to normal hearing and vision
* High-school educated
* Difficulty communicating in sentences, with some ability to use words independently

Exclusion Criteria:

* Severe apraxia of speech
* Other neurological conditions affecting communication (e.g., dementia)
* Uncontrolled psychiatric/psychological conditions affecting thinking and communication
* Active alcohol/substance abuse

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Production of target sentences on action description pictures | From baseline up to 1-week post training or 2-month post treatment
  Production accuracy (percent correct)
Comprehension of target sentences in a sentence-to-picture matching task | From baseline up to 1-week post training or 2-month post treatment
  Comprehension accuracy (percent correct)
Real-time comprehension of target sentences in a sentence-to-picture matching task | From baseline up to 1-week post training or 2-month post treatment
  Changes in eye fixations to the target picture

SECONDARY OUTCOMES:
Production of untrained sentences | From baseline up to 2-month post treatment
  Production accuracy (percent correct)
Connected speech production - story retell | From baseline up to 2-month post treatment
  Increased production of complex utterances as measured by proportion of sentence-level utterances out of all utterances
Connected speech production - picture description | From baseline up to 2-month post treatment
  Increased production of complex utterances as measured by proportion of sentence-level utterances out of all utterances

CONTACTS AND LOCATIONS:
Overall Officials: Jiyeon Lee, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual data with other researchers upon request. Other study materials (e.g., analytic code) will be made available via Open Science Forum. We will also make study-specific data and materials available for journal publications as supplemental materials, as relevant.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Researchers of OSF will access the study materials or data made available via OSF. Deidentified individual data can also be shared with other researchers upon requests and the PI will review each request. Other supporting materials such as study stimuli or protocols will be shared with other researchers upon request.